CLINICAL TRIAL: NCT06916936
Title: Effect of Peanut Butter on Gut and Metabolic Health in School-Aged Children
Brief Title: Effect of Peanut Butter on Gut and Metabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: The Peanut Institute (Other)
Responsible Party: Principal Investigator, Ravi Nagpal, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00005388; FA0000072215 (Other: Peanut Institute)
Record Dates: First submitted 2025-03-26; First posted 2025-04-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Dysbiosis
Keywords: microbiome; gut; nuts; peanut butter; metabolic health; dysbiosis; metagenomic; sleep quality; prebiotic; children
MeSH Terms: conditions — Dysbiosis; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut Butter Condition (Experimental): Peanut Butter (PB) Group: This condition involves a normal diet supplemented daily with a personalized portion of smooth peanut butter (Creamy Richards 100% Peanuts! Creamy Natural Peanut Butter) sandwiched between two plain unsalted saltine crackers (Unsalted Tops Premium Saltine Crackers). There is a limit of 16g of peanut butter per two crackers. The quantity of peanut butter provided daily will be equivalent to 20% of each participant's individual daily caloric intake. These caloric needs will be established using Dietary Guidelines for Americans (DGA) based on the participant's age and gender.
  Interventions: Other: Creamy Richards 100% Peanuts! Creamy Natural Peanut Butter
- Control Snack Condition (Active Comparator): Control (CTL) Group: This condition includes a normal diet supplemented daily with an isocaloric amount of a nut-free, vegetable oil-based chocolate spread (Cadbury Milk Chocolate) also sandwiched between two plain unsalted saltine crackers (Unsalted Tops Premium Saltine Crackers), with the same 16g limit per two crackers. The quantity of chocolate spread provided daily will be equivalent to 20% of each participant's individual daily caloric intake. These caloric needs will be established using Dietary Guidelines for Americans (DGA) based on the participant's age and gender
  Interventions: Other: Cadbury Milk Chocolate Spread

INTERVENTIONS:
Other: Creamy Richards 100% Peanuts! Creamy Natural Peanut Butter — Peanut Butter (PB) Group: Participants in this group will receive a daily snack consisting of a personalized portion of smooth peanut butter ("Creamy Richards 100% Peanuts! Creamy Natural Peanut Butter") spread between two plain unsalted saltine crackers ("Unsalted Tops Premium Saltine Crackers"). The amount of peanut butter will be limited to 16g per two crackers, but additional crackers will be provided if the personalized portion exceeds this limit
  Arms: Peanut Butter Condition
Other: Cadbury Milk Chocolate Spread — Control (CTL) Group: Participants in this group will receive a daily snack consisting of an isocaloric amount of a nut-free, vegetable oil-based chocolate spread ("Cadbury Milk Chocolate") spread between two plain unsalted saltine crackers ("Unsalted Tops Premium Saltine Crackers"). Similar to the peanut butter group, the chocolate spread will be limited to 16g per two crackers, with additional crackers provided if needed.
  Other Names: Control Snack; CTL; Isocaloric Spread
  Arms: Control Snack Condition

SUMMARY:
The goal of this is parallel arm, randomized clinical trial is to learn and understand the effect of daily smooth peanut butter consumption on gut and metabolic health of children age 6-13. The main objectives are:

Primary Objective: To determine the prebiotic effect of daily smooth peanut butter consumption for eight weeks on gut health, including microbiome-metabolome arrays, gut epithelial/barrier function, and gut transit time, in school-aged children.

Secondary Objective(s)

1. To determine the effect of daily smooth peanut butter consumption for eight weeks on metabolic and inflammatory health markers, and measures of sleep quality in school-aged children.
2. To determine the potential mechanisms and feasibility of incorporating peanut butter into the diets of school-aged children as part of healthy, personalized nutrition.

Research Intervention(s): Researchers compare two groups to see if there really is an effect of daily smooth peanut butter intake on gut and metabolic health. The two groups are:

1. The 1st condition (PB) includes a normal diet supplemented daily with personalized portion of smooth PB, sandwiched between two plain unsalted saltine crackers.
2. The 2nd condition (CTL) includes a normal diet supplemented daily with an isocaloric amount of a nut-free, vegetable oil-based chocolate spread, sandwiched between two plain unsalted saltine crackers.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in elementary or middle school (grades 1-8)
* Aged 6-13 years old
* Ability to speak and read in English

Exclusion Criteria:

* Intake of antibiotics in the last 3 months
* Intake of pre/pro/postbiotics in the last 3 months
* Food allergy to study foods

  * Any allergy to nuts or peanuts
* Any allergy to the isocaloric snack (chocolate or wheat)
* Regular consumption of nuts or peanuts greater than 2 servings / week
* Gastrointestinal disease (ulcerative colitis, Crohn's disease, diverticulosis, peptic ulcers, small intestinal bacterial overgrowth, short bowel syndrome, irritable bowel syndrome, gastroesophageal reflux disease), neurological (multiple sclerosis, meningitis, recent stroke) or endocrine disorders (uncontrolled thyroid disorders, growth hormone disorders, adrenal gland disorders, uncontrolled diabetes - A1C > 9%).
* Known to be pregnant (self-disclosed)

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Gut Microbiome Diversity | Baseline (day 0) Midpoint (week 4), and endpoint (week 8)
  Collected fecal samples will be used to determine microbiome profiles, including diversity and composition of bacteria.
Change in Oral Microbiome Diversity | Baseline (day 0), Endpoint (week 8)
  Oral swab samples are collected to determine oral diversity and composition of bacteria in the mouth before and after intervention.
Change in Fecal Metabolome | Baseline (day 0) and Endpoint (week 8)
  The endpoint of fecal metabolomics will be assessed by collecting fecal samples from participants at the beginning and end of the study. These samples will be analyzed using advanced techniques, such as mass spectrometry, to identify and quantify various metabolites present in the feces. The changes in the levels of specific metabolites, which can reflect shifts in gut microbiome composition and metabolic health, will be compared between pre- and post-intervention periods. This analysis will help determine how regular peanut butter intake affects metabolic processes and gut health.
Change in Serum Metabolome | Baseline (day 0), and Endpoint (week 8).
  The endpoint of serum metabolomics will be assessed by collecting blood serum from participants at the beginning and end of the study. These samples will be analyzed using advanced techniques, such as mass spectrometry, to identify and quantify various metabolites present in the serum. The changes in the levels of specific metabolites, which can reflect shifts in gut microbiome composition and metabolic health, will be compared between pre- and post-intervention periods. This analysis will help determine how regular peanut butter intake affects metabolic processes and gut health.

SECONDARY OUTCOMES:
Change in Gut Transit Time | Baseline (day 0), and endpoint (week 8)
  Evaluate changes in gut transit time after peanut butter or control snack consumption from baseline to final analysis, using a blue-dye capsule.
Change in Waist / Hip Circumference | baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in waist and hip circumference (centimeters), as well as waist-hip ratio at each study visit before, after and during peanut butter consumption, compared to a control snack.
Change in Habitual Dietary Intake | baseline (day 0), midpoint (week 4) and endpoint (week 8).
  Assess changes in habitual dietary intake via 3-day food logs, analyzed using nutrient analysis software (NDSR).
Change in Body Weight | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  the endpoint of body weight (kg) will be measured at each visit to assess changes in weight before and after 8 week consumption peanut butter or a control snack spread.
Change in Urinary Melatonin | Baseline (day 0) Midpoint (week 4), endpoint (week 8).
  Changes in melatonin (urine metabolite 6-sulphatoxymelatonin) will be assessed before, during and after 8-week consumption of peanut butter or control snack spread.
Change in Urinary Serotonin | Baseline (day 0) Midpoint (week 4), endpoint (week 8).
  Changes in urinary serotonin (urine metabolite 5-HIAA) will be assessed before, during and after 8-week consumption of peanut butter or control snack spread.
Change in Body Fat Percentage | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in body composition, including fat mass, expressed as a percentage of total weight (%). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during peanut butter or control snack consumption.
Change in Lipid Profiles | Baseline (day 0), endpoint (week 8)
  Relevant biomarkers are to be collected via venous blood samples to determine changes in cardiometabolic health including HDL, LDL, total cholesterol, and triglycerides. All will be expressed in units of mg/dL.
Change in Biomarkers of Inflammation | Baseline (day 0), Endpoint (week 8)
  Relevant biomarkers are to be collected via venous blood samples to determine changes in inflammation, including but not limited to C-reactive protein (CRP), IL-1 (Interleukin-1), IL-1 beta, IL-6, IL-10, IL-17, IL-23, Tumor Necrosis Factor Alpha (TNF-a), Interferon-gamma (IFN-Y). All will be expressed in units of pg/mL.
Change in Biomarkers of Intestinal Barrier Function | Baseline (day 0), endpoint (week 8).
  Relevant biomarkers are to be collected via venous blood samples to determine changes in intestinal barrier function including LPS (lipopolysaccharides), LBP (lipopolysaccharide binding protein), CD14, Secretory IgA. All will be expressed in units of pg/mL.
Change in Lean Mass | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in body composition, including lean mass (kg). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during peanut butter or control snack consumption.
Change in Biomarkers of Appetite | baseline (day 0), endpoint (week 8)
  Relevant biomarkers are to be collected via venous blood samples to determine changes in appetite including Insulin, Glucagon, glucagon-like peptide 1 (GLP-1), Adiponectin, Leptin, Ghrelin, and Peptide YY. All will be expressed in units of pg/mL.
Change in Rested, Seated Blood Pressure | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  This outcome measure will measure changes in blood pressure taken at rest in the seated position at each visit, before during and after peanut butter or control snack consumption, expressed as systolic over diastolic blood pressure in units of millimeters of mercury (mmHg).
Change in Fasting Blood Glucose | Baseline (day 0), endpoint (week 8).
  Venous blood samples will be collected to determine changes in fasting blood glucose (expressed as mg/DL).
Dietary Adherence | Daily, baseline through endpoint (week 8)
  Assess adherence to the intervention and control snack throughout the study, as determined by dietary adherence logs kept by the participants each week. Adherence is expressed as a daily percent (%) consumption of their assigned snack
Change in Total Body Water | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in body composition, including, total body water (L). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during peanut butter or control snack consumption.
Change in Intracellular Fluid | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in body composition, including intracellular fluid (L). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during peanut butter or control snack consumption.
Change in Extracellular Fluid | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in body composition, including extracellular fluid (L). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during peanut butter or control snack consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Nagpal, Ph.D., Principal Investigator — Florida State University
Locations (1):
- Florida State Univresity - The Gut Biome Lab, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified IPD will not be retain past three years, at the time of this submission the researchers does not plan to make IPD available

REFERENCES:
- See also: The corresponding official Gut Biome Lab website is linked here — https://thegutbiomelab.annescollege.fsu.edu/